CLINICAL TRIAL: NCT06831708
Title: A Randomized Controlled Trial Comparing Short-Term Psychoanalytic Therapy and Cognitive Behavioral Therapy for Generalized Anxiety Disorder
Brief Title: RCT of Short-Term Psychoanalytic vs. Cognitive Behavioral Therapy for GAD
Acronym: (RCT-GAD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beykoz University (Other)
Collaborators: Uskudar University (Other); Istanbul Nisantasi University (Other)
Responsible Party: Principal Investigator, Eda Yilmazer, Principle Investigator, Beykoz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Beykoz Psychoanalysis vs CBT
Record Dates: First submitted 2025-02-01; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder; Psychoanalytic Therapy; Cognitive Behavioral Therapy; RCT; Anxiety; Short-Term Psychotherapy
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into one of three parallel arms: a psychoanalytic therapy arm, a CBT arm, or a control (waiting list) arm. Each arm will consist of 20 participants, with interventions delivered over 12 weekly sessions.
Masking Description: There is no masking in this study. All participants and study personnel will be aware of the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Psychoanalytic Therapy (Experimental): Participants in this arm will receive short-term psychoanalytic therapy delivered via a standardized framework. Although the approach is not strictly manualized, a set of core principles (including exploration of unconscious conflicts, transference, and resistance) will guide therapy. The therapy will be administered in 12 weekly sessions, each lasting 50 minutes, by two of the study authors trained in this approach.
  Interventions: Behavioral: Psychoanalytic Psychotherapy
- Cognitive Behavioral Therapy (CBT) (Experimental): Participants in this arm will receive a structured, manualized cognitive behavioral therapy (CBT) intervention specifically designed for the treatment of Generalized Anxiety Disorder (GAD). Therapy will consist of 12 weekly sessions, each 50 minutes in duration, delivered by two of the study authors with specialized CBT training.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Control (Waiting List) (No Intervention): Participants in this arm will be placed on a waiting list for treatment. They will not receive any active psychotherapeutic intervention during the study period but may continue any standard care they are already receiving.

INTERVENTIONS:
Behavioral: Psychoanalytic Psychotherapy — This intervention involves short-term psychoanalytic therapy based on a standardized framework. Although not rigidly manualized, the treatment protocol includes core psychoanalytic concepts (such as transference, resistance, and the exploration of unconscious conflicts). Sessions will be conducted weekly (50 minutes each) for a total of 12 sessions. This intervention is delivered by two study authors who have undergone dedicated training and calibration to ensure consistent application of the framework.
  Arms: Psychoanalytic Therapy
Behavioral: Cognitive Behavioral Therapy (CBT) — This intervention consists of a structured and manualized CBT program specifically tailored for individuals with Generalized Anxiety Disorder (GAD). The intervention includes defined session objectives, cognitive restructuring techniques, behavioral experiments, and homework assignments. Participants will receive 12 weekly sessions (50 minutes each), delivered by two study authors who are trained in CBT.
  Arms: Cognitive Behavioral Therapy (CBT)

SUMMARY:
This study is a randomized controlled trial designed to compare the effectiveness of two types of short-term psychotherapy-psychoanalytic therapy and Cognitive Behavioral Therapy (CBT)-in treating Generalized Anxiety Disorder (GAD). A total of 60 adult participants with a confirmed diagnosis of GAD will be enrolled and randomly assigned to one of three groups: one group will receive psychoanalytic therapy, a second group will receive CBT, and a third group will serve as a control (waiting list) group. Each treatment group will participate in 12 weekly sessions, with each session lasting 50 minutes.

In the psychoanalytic therapy group, therapy will follow a standardized framework based on core psychoanalytic principles such as exploring unconscious conflicts, transference, and resistance. While this approach is flexible, all therapists will be trained and calibrated to apply these core principles consistently. In contrast, the Cognitive Behavioral Therapy (CBT) group will receive a structured, manualized intervention specifically designed for Generalized Anxiety Disorder (GAD). The control group will not receive any active psychotherapy during the study period but will continue to receive any standard care they are already using.

The primary outcome of the study will be the change in anxiety symptoms measured by the Beck Anxiety Inventory (BAI) from before treatment to after the 12 sessions. Secondary outcomes will include measures of quality of life (using the World Health Organization Quality of Life Instrument [WHOQOL-BREF]), depressive symptoms (using the Beck Depression Inventory-II [BDI-II]), functional impairment (using the World Health Organization Disability Assessment Schedule II [WHODAS II]), the quality of the therapeutic relationship (using the Working Alliance Inventory [WAI]), and overall treatment satisfaction.

The study is designed to be completed within a six-month period: one month for recruitment, one month for baseline assessments and clinical checks, and three months for the intervention. Data will be collected at baseline and immediately after the intervention, with the goal of analyzing and publishing the results as soon as possible following treatment completion. This study has received ethical approval from the Üsküdar University Ethics Committee and is intended to inform future research on effective treatments for Generalized Anxiety Disorder (GAD).

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) is designed to rigorously compare the clinical outcomes of two psychotherapeutic interventions for Generalized Anxiety Disorder (GAD)-short-term psychoanalytic therapy and Cognitive Behavioral Therapy (CBT)-against a control (waiting list) condition. The study will be conducted at a single center with a total sample of 60 participants who have been diagnosed with GAD according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria within the past two years. Participants will be stratified and randomly assigned in equal numbers (n=20 per group) to one of the three study arms.

Intervention Details:

Psychoanalytic Therapy Arm:

Although psychoanalytic therapy is inherently flexible and individualized, for the purposes of this study a standardized framework will be employed. This framework is based on core psychoanalytic principles such as the exploration of unconscious conflicts, the dynamics of transference, and the management of resistance. The approach is not rigidly manualized; instead, it is standardized through:

Pre-intervention Training: Therapists will engage in specific training sessions to discuss and agree on key therapeutic elements and session structure.

Calibration Meetings: Regular meetings will be held to ensure consistent application of the framework.

Fidelity Monitoring: A session checklist will be utilized to document the presence of core components in each session. Selected sessions may be recorded (with participant consent) for review by an independent clinician to ensure adherence to the agreed-upon framework.

Cognitive Behavioral Therapy (CBT) Arm:

The CBT intervention will follow a structured, manualized protocol tailored specifically for treating GAD. This intervention includes:

Manualized Sessions: Each of the 12 weekly sessions (50 minutes each) will have defined objectives, cognitive restructuring techniques, behavioral experiments, and homework assignments.

Standardization and Supervision: Therapists will receive training in the manualized approach and undergo regular supervision, including periodic review of session recordings and fidelity checklists to ensure strict adherence to the protocol.

Control Arm:

Participants in the control group will be placed on a waiting list for treatment. They will not receive any active psychotherapeutic intervention during the study period, although they may continue any ongoing standard care. This group is included to control for the effects of time and natural fluctuations in anxiety symptoms.

Assessment and Outcome Measures:

Data will be collected at two time points: at baseline (prior to the start of the intervention) and immediately following the completion of the 12-week intervention phase. The primary outcome measure is the change in anxiety symptoms as assessed by the Beck Anxiety Inventory (BAI). Secondary outcomes include:

Quality of Life: Measured by the World Health Organization Quality of Life Instrument (WHOQOL-BREF).

Depressive Symptoms: Measured by the Beck Depression Inventory-II (BDI-II). Functional Impairment: Assessed using the World Health Organization Disability Assessment Schedule II (WHODAS II).

Therapeutic Alliance: Evaluated via the Working Alliance Inventory (WAI), administered after the third session.

Treatment Satisfaction: Assessed through a post-treatment satisfaction questionnaire.

Study Timeline:

Recruitment Period: Approximately one month will be dedicated to recruiting the required sample.

Baseline Assessment and Clinical Evaluation: A subsequent one-month period will be used to perform baseline assessments, including a clinical evaluation by a collaborating psychiatrist.

Intervention Phase: Over the next three months, participants will undergo 12 weekly therapy sessions.

Post-Treatment Evaluation: Data collection for outcome measures will occur immediately following the intervention, allowing for timely analysis and dissemination of results.

Data Handling and Analysis:

Data collection will be executed using secure online platforms for questionnaires and standardized assessment tools. Clinical evaluations may be conducted in-person or via secure video conferencing, ensuring flexibility and participant convenience. All data will be anonymized and stored in compliance with current data protection regulations.

The statistical analysis will primarily focus on changes in Beck Anxiety Inventory (BAI) scores using Analysis of Variance (ANOVA) or repeated measures ANOVA to compare the effects between the three groups. Secondary outcome measures will be analyzed similarly. An intention-to-treat (ITT) analysis will be applied, including all participants randomized to the study, to preserve the benefits of randomization and reduce bias. Data analysis will be carried out using validated statistical software packages such as Statistical Package for the Social Sciences (SPSS) or R.

Ethical and Administrative Considerations:

The study has received ethical approval from the Üsküdar University Ethics Committee. Written informed consent will be obtained from all participants prior to enrollment. The study has been designed with strict adherence to ethical standards to ensure participant safety, confidentiality, and data integrity.

This protocol has been structured to enable rapid completion of the study within a six-month period while providing robust and reliable data. The outcomes of this study are expected to inform clinical practice by clarifying the comparative effectiveness of a structured Cognitive Behavioral Therapy (CBT) intervention versus a standardized framework for psychoanalytic therapy in the treatment of Generalized Anxiety Disorder (GAD). Future studies may extend these findings by including longer follow-up periods to assess the durability of therapeutic effects.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* A confirmed diagnosis of Generalized Anxiety Disorder (GAD) according to DSM-5 criteria, with the diagnosis made within the past 2 years.
* No participation in any form of psychotherapy during the past 6 months.
* Ability and willingness to attend 12 weekly therapy sessions (50 minutes each) over the 3-month intervention period.
* For participants receiving online sessions: access to a stable internet connection and the necessary technology.
* Ability to understand and provide written informed consent.

Exclusion Criteria:

* Presence of significant comorbid psychiatric disorders that could interfere with participation or assessment (e.g., bipolar disorder, psychotic disorders, substance use disorders, eating disorders).
* Recent changes in psychotropic medication (i.e., medication changes within the past 3 months, unless on a stable dose).
* Severe medical or neurological conditions that may interfere with study participation or data interpretation.
* Current participation in another clinical trial or structured psychotherapy program.
* Any condition that, in the opinion of the investigators, would compromise the safety or compliance of the participant in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Beck Anxiety Inventory (BAI) | Baseline (pre-treatment) and immediately post-treatment (after completion of 12 weekly sessions, approximately 3 months after baseline)
  The primary outcome is the change in anxiety severity measured by the Beck Anxiety Inventory (BAI), a 21-item self-report scale rated from 0 ("Not at all") to 3 ("Severely"). Total scores range from 0 to 63, with higher scores indicating greater anxiety severity: 0-7 (minimal), 8-15 (mild), 16-25 (moderate), and 26-63 (severe). The BAI will be administered at baseline and after 12 weekly sessions. The primary analysis will compare changes in BAI scores across the three study arms (psychoanalytic therapy, Cognitive Behavioral Therapy [CBT], and control) to assess treatment efficacy for Generalized Anxiety Disorder (GAD).

SECONDARY OUTCOMES:
World Health Organization Quality of Life (WHOQOL-BREF Score) | Baseline (pre-treatment) and Immediately Post-Treatment (after 12 sessions, approximately 3 months after baseline)
  The WHOQOL-BREF is a 26-item self-report questionnaire assessing quality of life across four domains: physical health, psychological health, social relationships, and environment. Each item is rated on a 5-point Likert scale, with higher scores indicating better quality of life. Domain scores range from 4 to 20 and can be transformed to a 0-100 scale. The WHOQOL-BREF will be administered at baseline and post-intervention to assess treatment impact on quality of life in individuals with Generalized Anxiety Disorder (GAD).
Beck Depression Inventory (BDI-II Score) | Baseline (pre-treatment) and Immediately Post-Treatment (after 12 sessions)
  The BDI-II is a 21-item self-report questionnaire assessing depressive symptom severity over the past two weeks. Each item is rated from 0 to 3, with total scores ranging from 0 to 63 (higher scores indicating more severe depression): 0-13 (minimal), 14-19 (mild), 20-28 (moderate), 29-63 (severe). The BDI-II will be administered at baseline and post-treatment to assess changes in depressive symptoms in participants with Generalized Anxiety Disorder (GAD).
World Health Organization Disability Assessment Schedule II (WHODAS II Score) | Baseline (pre-treatment) and Immediately Post-Treatment (after 12 sessions)
  The WHODAS II is a 36-item questionnaire assessing functioning across six domains: cognition, mobility, self-care, getting along, life activities, and participation. Each item is rated on a 5-point scale, with total scores ranging from 0 (no disability) to 100 (full disability). Higher scores indicate greater functional impairment. The WHODAS II will be administered at baseline and post-treatment to assess changes in daily functioning and disability levels.
The Working Alliance Inventory (WAI Score) | Baseline (pre-treatment) and Immediately Post-Treatment (after 12 sessions)
  The WAI is a self-report questionnaire assessing the therapeutic relationship across three components: goal agreement, task consensus, and bond development. The original 36-item WAI uses a 7-point scale (1 = never, 7 = always), with higher scores indicating a stronger alliance. The 12-item WAI-Short Form (WAI-S) is often used in clinical settings. The WAI will be administered after the third session to assess the therapeutic relationship's role in treatment outcomes for Generalized Anxiety Disorder (GAD).

CONTACTS AND LOCATIONS:
Overall Officials: Eda Yılmazer, Phd, Principal Investigator — Beykoz University; Metin Çınaroğlu, Phd, Principal Investigator — Istanbul Nisantasi University
Locations (1):
- Beykoz University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
We plan to share de-identified individual participant data (IPD) collected in this study. The shared data will include the raw outcome measures (e.g., Beck Anxiety Inventory, WHOQOL-BREF, Beck Depression Inventory-II, WHODAS II, Working Alliance Inventory, and treatment satisfaction scores), baseline demographic information, and clinical assessment data. Supporting documentation-including the study protocol, statistical analysis plan (SAP), informed consent form (ICF), clinical study report (CSR), and analytic code-will also be provided to facilitate secondary analyses. No identifying information will be shared.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: IPD and supporting documents will be made available beginning 6 months after publication of the primary manuscript in a peer-reviewed journal and will remain available for a period of 5 years thereafter.
Access Criteria: Access to the IPD and supporting documentation will be granted to qualified researchers who submit a methodologically sound research proposal. Data will be provided through a secure data access portal following review and approval by the study team. Researchers will be required to sign a data use agreement to ensure the data are used solely for research purposes and in compliance with applicable privacy regulations.